CLINICAL TRIAL: NCT03223779
Title: Phase Ib/II Study of TAS-102 Plus Radiation Therapy for the Treatment of the Liver in Patients With Hepatic Metastases From Colorectal Cancer
Brief Title: Study of TAS-102 Plus Radiation Therapy for the Treatment of the Liver in Patients With Hepatic Metastases From Colorectal Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Taiho Oncology, Inc. (Industry)
Responsible Party: Principal Investigator, Jennifer Wo, Director, Gastrointestinal Service, Department of Radiation Oncology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-231
Record Dates: First submitted 2017-07-12; First posted 2017-07-21 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — trifluridine tipiracil drug combination; Trifluridine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- TAS-102 (Experimental): * Photon treatments will be performed on a linear accelerator
  * Photon SBRT will be given during TAS-102 dosing
  * TAS-102 dosing occurs on days 1 through 5 and 8 through 12
  * TAS-102 tablets should be taken twice a day orally
  Interventions: Drug: TAS-102; Radiation: Photon SBRT

INTERVENTIONS:
Drug: TAS-102 — Trifluridine stops DNA replication which may prevent the cancer cells from growing
  Other Names: Lonsurf; Trifluridine
Radiation: Photon SBRT — SBRT stands for Stereotactic Body Radiation Therapy. Radiation may help to kill the cancer cells while protecting your normal tissue cells

SUMMARY:
This research study is studying a drug in combination with radiation therapy as a possible treatment for hepatic metastases from colorectal cancer.

The interventions involved in this study are:

* Trifluridine (TAS-102)
* Radiation Therapy

DETAILED DESCRIPTION:
This is a Phase I/II clinical trial. Patients are being asked to participate in the Phase I portion of the study. A Phase I clinical trial tests the safety of an investigational intervention and also tries to define the appropriate dose of the investigational drug to use for further studies. "Investigational" means that the intervention is being studied.

The FDA (the U.S. Food and Drug Administration) has approved Trifluridine as a treatment option for this disease.

The FDA has not approved Trifluridine in combination with radiation therapy as a treatment option for this disease.

In this research study, the investigators are determining the safest and most effective dose of Trifluridine in combination with radiation therapy in participants with hepatic metastases from colorectal cancer.

Trifluridine stops DNA replication which may prevent the cancer cells from growing. Radiation may help to kill the cancer cells while protecting normal tissue cells. Studies have shown Trifluridine may make radiation more effective.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have biopsy-proven diagnosis of a colorectal cancer with 1-4 liver metastases. There is no upper size limit and participants must have at least 800 mL of uninvolved liver. Liver metastases may be diagnosed by imaging alone, no liver biopsy is required. Extrahepatic disease is allowed if 1) it has been stable for 3 months prior to study entry, 2) the dominant disease burden is intrahepatic and 3) the patient is referred for definitive radiation therapy to the disease in the liver.
* Participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 10 mm with spiral CT scan. See Section 13 for the evaluation of measurable disease.
* Participants may have had prior chemotherapy, targeted biological therapy (i.e. sorafenib), surgery, transarterial chemoembolization (TACE), radiofrequency ablation, or cryosurgery for their disease as long as the prior therapy occurred more than 3 weeks before the first radiation treatment. Patients may not have had prior liver directed radiation, including radioembolization.
* Participants must be 18 years of age or older.
* Because no dosing or adverse event data are currently available on the use of high dose liver radiation in participants <18 years of age, children are excluded from this study.
* Expected survival must be greater than three months.
* ECOG Performance Status 0 or 1..
* Participants must have liver metastases deemed unresectable due to anatomy, medical fitness, or presence of extrahepatic disease.
* Participants must have normal organ and marrow function as defined below. History of transfusion is acceptable and transfusions may be given to meet eligibility requirements.

  * Hgb ≥ 9g/dL
  * Absolute neutrophil count ≥ 1,500/mm3
  * Platelets ≥ 75,000/mm3
  * Total bilirubin ≤ 1.5 X institutional upper limit of normal
  * AST (SGOT) and ALT (SGPT) ≤ 1.5 X institutional upper limit of normal
  * Creatinine ≤ 1.5 mg/dl or creatinine clearance ≥ 60 mL/min/1.73 m2 (Calculated per Cockroft & Gault formula) for subjects with creatinine levels above institutional normal.
* If patient has underlying cirrhosis, only Child-Pugh classification Group A patients should be included in this study. Clinical assessment of ascites and encephalopathy is required. Child-Pugh classification must be determined for all study participants at the time of eligibility analysis. As albumin and PT/INR are required for Child-Pugh classification; these labs should be drawn with other labs required for eligibility analysis. See Appendix B for Child-Pugh classification table.
* The effects of radiation on the developing human fetus are known to be teratogenic and the safety of TAS-102 in pregnant women and their fetuses has not been established. Therefore, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 6 months after stopping study treatment. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.
* Ability to take oral medications (i.e. no feeding tube and able to swallow whole)

Exclusion Criteria:

* Women who are pregnant or lactating. Patients must be either surgically sterile (via hysterectomy or bilateral tubal ligation), post menopausal or using acceptable methods of contraception if they are of child bearing potential. Female patients of child bearing potential must have a negative serum or urine pregnancy test within 7 days prior to starting drug. Because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with radiation, breastfeeding should be discontinued if the mother is treated with radiation.
* Participants with gross ascites or encephalopathy
* Participants with local conditions or systemic illnesses that would reduce the local tolerance to radiation treatment, such as serious local injuries, active collagen vascular disease, etc.
* Participants who have had prior liver directed radiation treatment, including selective internal radiation (SIRspheres or Theraspheres)
* Participants with a serious medical illness that may limit survival to less than 3 months
* Participants who have had chemotherapy or radiotherapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C) prior to starting study treatment or those who have not recovered from adverse events due to agents administered more than 3 weeks earlier.
* Participants who are receiving any other investigational agents, or any other anti-cancer therapy during study treatment.
* Participants with any uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or serious psychiatric illness/social situations that would limit compliance with study requirements.
* Participants who have previously received TAS-102

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-10-13 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | From start of treatment until 4 weeks after the end of treatment
  MTD will be determined using a 3 + 3 dose escalation. 3 participants enrolled at the starting dose of 20 mg/m2 BID (Bis in die, Latin for twice daily). Based on the number of dose limiting toxicities (DLT), the dose can be either be increased to 25 mg/m2 BID then 30 mg/m2 BID or it could be reduced to 15 mg/m2 BID.
  * If 0 out of 3 have DLT, enroll 3 participants at next dose level
  * If ≥ 2 DLT out of 3 or 6 participants in a dose cohort have DLT, this will be the MTD and 3 additional participants are enrolled at next lowest dose if only 3 were treated at that level so far.
  * If 1 out of 3 have DLT, 3 more enrolled at current dose level. If no DLT in those 3, move to next dose level. If ≥ 1 DLT, declare this the MTD and enroll 3 additional at next lowest dose if only 3 treated so far.
  * If ≤ 1 out of 6 DLT at highest dose level below maximally administered dose, MTD is generally the rerecorded phase 2 dose (RP2D). Dose level 3 is RP2D if MTD not reached.
The Duration of Local Control | Baseline, 1 month post treatment, every 6 months for two years or until death
  Local control is the absence of local failure defined as evidence of tumor growth/regrowth that meets Response Evaluation Criteria In Solid Tumors (RECIST) criteria for progressive disease in any direction beyond that present in pre-treatment imaging studies of the treated lesion(s). The duration of local control will be measured from the start date of protocol treatment until the date of local failure.
  * Marginal failure is defined as appearance of tumor growth at the margin of the target volume.
  * Nodal failure is defined as failure in regional lymph nodes (i.e. porta-hepatis, para-aortic, diaphragmatic).
  * Distant failure is defined as appearance of tumor at sites beyond marginal and regional nodal sites.
  * Intrahepatic recurrence is defined as any new lesion elsewhere in the liver and separate from local failure.

SECONDARY OUTCOMES:
Toxicity associated with TAS-102 combined with SBRT | From start of treatment until 4 weeks after the end of treatment
  Summary of the Adverse events experienced during treatment. Adverse events are assessed with Common Terminology Criteria for Adverse Events (CTCAE) 4.0.
Progression Free Survival | from the start of treatment until 2 years, or until time of progression/death
  Progression-free survival (PFS) will be measured from the start date of protocol treatment (first TAS-102 dose and/or first SBRT fraction) to the earlier date of first failure at any pre-treatment or new site (defined in 'Duration of Local Control' section) or death. PFS will be censored at the date of last follow-up for participants still alive who have not failed.
Overall Survival | from the start of treatment until 2 years, or until time of death
  Overall survival (OS) will be measured from the start date of protocol treatment (first TAS-102 dose and/or first SBRT fraction) to the date of death. OS will be censored at the date of last follow-up for participants who are still alive.
Association between KRAS or BRAF mutation status with local control | Baseline, 1 month post treatment, every 6 months for two years or until death
  Association between KRAS or BRAF mutation status with local control will be assessed using Gray's test with death as a competing risk in the absence of local failure. Local control is defined in the 'Duration of Local Control' description.
Serial ctDNA | Baseline, week 1, week 2, 1 month post treatment, at the time of progression
  Serial ctDNA will be analyzed by descriptive methods to identify potential trends and correlations with synchronous radiologic endpoints (baseline, one month post-treatment). ctDNA level (detectable versus negative) at early (week 1, week 2) and post-treatment (one month) assessments will be analyzed for differences in local control

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Y. Wo, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No